CLINICAL TRIAL: NCT07258017
Title: Multidimensional Impact Analysis of Interactive Video Health Intervention on Quality of Life and Clinical Rehabilitation Indicators in Patients With Early Postoperative Bowel Obstruction: A Randomized Controlled Tria
Brief Title: Impact of Interactive Video Health Intervention on Quality of Life After Bowel Obstruction Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changsha Fourth Hospital (Other Government)
Responsible Party: Principal Investigator, Li Zhang, Principal Investigator, Changsha Fourth Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSSDSYY-YXLL-SC-2024-02-20
Record Dates: First submitted 2025-09-24; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-01

CONDITIONS: Intestinal Obstruction; Postoperative Complications
MeSH Terms: conditions — Intestinal Obstruction; Postoperative Complications

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Care Control Group (Active Comparator)
  Interventions: Behavioral: Conventional care
- Interactive Video Health Intervention Group (Experimental)
  Interventions: Behavioral: Interactive Video Health Intervention

INTERVENTIONS:
Behavioral: Conventional care — Standard conventional care including condition monitoring, basic medical treatment (gastrointestinal decompression, fluid replacement, correction of water-electrolyte disorders), and non-structured health education. Represents the current standard of care for postoperative bowel obstruction patients without the additional video-based intervention component.
  Arms: Conventional Care Control Group
Behavioral: Interactive Video Health Intervention — A structured interactive video intervention consisting of 5 modular videos covering disease knowledge, rehabilitation exercises, and dietary guidance. The videos use animation demonstrations, case analyses, and expert explanations, with interactive elements such as Q&A sessions and polls. Initiated 24 hours post-surgery, patients can self-paced viewing using tablet devices with researcher support.
  Arms: Interactive Video Health Intervention Group

SUMMARY:
Objective: To investigate the multidimensional effects of an interactive video health intervention on the quality of life and clinical rehabilitation indicators of patients with early postoperative bowel obstruction.

Methods: The study consists of two phases. Phase 1 (January 2019-December 2020) involves the development and psychometric validation of a Postoperative Quality of Life Assessment Scale for Early Intestinal Obstruction, with approximately 150 patients. Phase 2 (January 2021-January 2025) is a randomized controlled trial enrolling about 310 eligible patients (aged 18-75 years, with basic cognitive ability, diagnosed with early postoperative bowel obstruction after abdominal surgery). Participants are randomly assigned to either a control group (conventional care, including condition monitoring, basic treatment, and non-structured health education) or a study group (conventional care plus an interactive video health intervention consisting of five modular videos covering disease knowledge, rehabilitation, and diet, initiated 24 hours post-surgery).

Primary and secondary outcomes will include quality of life (assessed with the validated scale), clinical rehabilitation indicators (such as obstruction relief time and hospitalization duration), electrogastrogram parameters, and gut microbiota diversity (16S rRNA sequencing).

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with early postoperative intestinal obstruction after abdominal surgery based on clinical symptoms, physical examination and imaging
* Aged between 18 and 75 years
* With basic cognitive ability and comprehension
* Informed consent obtained directly from patients; family members provided supplementary consent

Exclusion Criteria:

* Serious underlying diseases
* Serious mental diseases
* Audio-visual impairment that prevents normal reception of interactive video information
* Poor compliance

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 462 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2025-01-13 (Actual); Study Completion 2025-01-24 (Actual)

PRIMARY OUTCOMES:
Quality of Life (QoL) Score | Baseline (pre-intervention, within 24 hours after surgery) and at hospital discharge (average 8-10 days after randomization).
  Scale consists of multiple domains assessing physical, psychological, and social functioning. Scores range from 0 to 100, with higher scores indicating better quality of life.

SECONDARY OUTCOMES:
Time to Relief of Intestinal Obstruction | From randomization to hospital discharge (daily assessment, average 8-10 days)
  Time from randomization to relief of intestinal obstruction symptoms (abdominal pain, distension, and resumption of defecation/flatus), measured in hours using daily clinical evaluation and patient report.
Duration of Hospitalization | From the day of surgery through hospital discharge (an average of 7-10 days)
  Total number of days from the date of surgery to the date of hospital discharge, as recorded in hospital medical records. This indicator reflects postoperative recovery efficiency and the impact of the interactive video intervention on clinical outcomes.
Electrogastrogram (EGG) Parameters - Gastric Antrum Slow-Wave Amplitude | 24 hours post-intervention initiati
  Gastric antrum slow-wave amplitude measured in microvolts (μV) using electrogastrogram at specified time points.
Electrogastrogram (EGG) Parameters - Gastric Slow-Wave Frequency | 24 hours post-intervention initiation and
  Gastric slow-wave frequency measured in cycles per minute (cpm) using electrogastrogram at specified time points.
Title: Gut Microbiota Diversity (Shannon Index) | First postoperative defecation (typically 3-5 days post-surgery)
  Alpha diversity of gut microbiota measured by Shannon index using 16S rRNA sequencing of fecal samples.

OTHER OUTCOMES:
Postoperative Quality of Life Assessment Scale Validation - Reliability Metrics | At postoperative day 7 (single assessment after intervention)
  Internal consistency of the Postoperative Quality of Life Assessment Scale for Early Intestinal Obstruction, assessed using Cronbach's alpha (range 0-1; higher scores indicate better internal consistency).
Postoperative Quality of Life Assessment Scale Validation - Construct Validity Metrics | At postoperative day 7 (single assessment after intervention)
  Construct validity of the Postoperative Quality of Life Assessment Scale for Early Intestinal Obstruction (PQOL-EO), assessed using Average Variance Extracted (AVE) and Composite Reliability (CR). Both are unitless indices (range 0-1), where higher values indicate better construct validity and internal consistency of the scale.
Expert Consensus Agreement on Questionnaire Items | During the pre-intervention development phase (single assessment prior to participant enrollment)
  Percentage of questionnaire items rated as "appropriate" or "highly relevant" by an expert panel using a 5-point Likert scale (1 = not relevant to 5 = highly relevant). Higher scores indicate greater content validity and expert consensus regarding the Postoperative Quality of Life Assessment Scale for Early Intestinal Obstruction (PQOL-EO).

CONTACTS AND LOCATIONS:
Locations (1):
- The Fourth Hospital of Changsha, Changsha, Hunan, China

REFERENCES:
- [Derived] Yao L, Wu D, Liu J, Zhang X, Zhang L. Multidimensional impact analysis of interactive video health intervention on quality of life and clinical rehabilitation indicators in patients with early postoperative bowel obstruction: a randomized controlled trial. Int J Colorectal Dis. 2026 Jan 8;41(1):19. doi: 10.1007/s00384-025-05051-0. PMID 41507597